CLINICAL TRIAL: NCT02701088
Title: Phase II Study of SIB-IMRT in Combination With 5-FU and Mitomycin-C Among Patients With Locally Advanced Anal Canal Cancer: Efficacy, Safety and Quality of Life
Brief Title: Study of SIB-IMRT in Combination With 5-FU and Mitomycin-C Among Patients With Locally Advanced Anal Canal Cancer: Efficacy, Safety and Quality of Life
Acronym: CANAL-IMRT-01
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: Accuray Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CANAL-IMRT-01
Record Dates: First submitted 2015-12-23; First posted 2016-03-08 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced Anal Canal Cancer
MeSH Terms: interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Concomitant chemotherapy and radiotherapy (Experimental): Chemoradiotherapy with two cycles of 5FU and Mitomycin-C plus radiotherapy by SIB-IMRT (for simultaneous integrated boost intensity modulated radiation therapy) day 1 to day 50 in 36 fractions
  Interventions: Drug: 5Fluorouracile and Mitomycin-C; Radiation: Simultaneously integrated boost of intensity modulated radiation therapy (SIB-IMRT) by tomotherapy

INTERVENTIONS:
Drug: 5Fluorouracile and Mitomycin-C — All the patients will receive radiochemotherapy with two cycles of 5FU (1,000 mg/m²/d with 96-h infusion, days 1-5 and 29-33 of SIB-IMRT) and Mitomycin-C (10 mg/m², days 1 and 29).
Radiation: Simultaneously integrated boost of intensity modulated radiation therapy (SIB-IMRT) by tomotherapy — SIB-IMRT schedule of 61.2 Gy/1.7 Gy to the primary tumor, 57.60 Gy / 1.6 Gy to involved nodes, and 54 / 1.5 Gy to elective pelvic lymph nodes.

SUMMARY:
Anal canal carcinoma (ACC) represents 1.2% of digestive cancers. Its incidence is increasing. As epidermoid ACC (95% of ACC) are particularly sensitive to radio and chemotherapy, concomitant radio-chemotherapy is the standard treatment of locally advanced ACC, with proven efficacy on locoregional control, anal sphincter preservation, progression-free survival and complete response rate higher than 80%.

Nevertheless, conventional radiotherapy frequently induces significant non-haematological toxicities requiring treatment interruptions. Thus, treatment usually includes a chemotherapy (5-Fluorouracil and Mitomycine-C) and 25 fractions of 1.8 Gy followed by a planned 1-week (or more) interruption and a boost, for a total 54-60 Gy radiation dose over 9 weeks.

Considering the numerous anatomic pelvic structures, ACC has become a localisation of interest for Intensity-Modulated Radiation Therapy (IMRT) associated with less toxicity.

However, IMRT induces grade≥3 cutaneous toxicities requiring irradiation breaks. Dose escalade did not show its interest: 60 Grays remains the standard.

Assuming the deleterious effect of increased overall treatment time on local control and survival in head-and-neck and cervical cancers and the epidermoid histology of ACC, the benefit of no irradiation break on ACC tumour control is of interest.

IMRT offers the possibility to deliver different doses to different target volumes simultaneously by altered fractionation schedule like SIB-IMRT (simultaneously integrated boost-IMRT). Several SIB-IMRT schedules have been retrospectively evaluated. Similar results were observed with moderate doses and schedules delivering higher doses with short interruptions. Nevertheless, standard SIB-IMRT schedule in ACC still not exist.

ELIGIBILITY:
Inclusion Criteria:

* WHO performance status ≤ 2
* Age > 18 years
* Epidermoid anal canal carcinoma histologically proven, locally advanced with an indication of radiation of pelvic and inguinal nodes concomitantly to chemotherapy
* The T corresponds to the larger dimension of tumor at the rectal examination and the N is assessed by imaging pelvic MRI-imaging, CT-scan, optionally PET-CT). Eligible tumors are: T2 more than 4 cm N0-N3, T2-T4 N1-N3 or usN1, T3-T4 N0, M0 according to the 6th edition of the American Joint Committee on cancer staging manual.
* Laboratory data obtained ≤ 14 days prior to registration on study, with adequate bone marrow, hepatic and renal function defined as follows: hemoglobinemia, neutrophil, platelet counts, bilirubin and creatinin level
* Informed consent form

Exclusion Criteria:

* Previous invasive cancer within 5 years except basocellular cancer and in situ cervical cancer
* Tumors with predominant skin involvement
* Presence of metastases
* History of pelvic irradiation
* Contraindication to radiotherapy or chemotherapy
* Known HIV positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy: The 3-month locoregional control rate | 3 months after the end of radiotherapy
  The 3-month locoregional control rate after the end of IMRT by helical tomotherapy defined by the proportion of patients alive with no local disease progression 3 months after the end of radiotherapy
Tolerance profile: Proportion of patients with no significant toxicities responsible for irradiation breaks | Until 11 weeks after treatment start
  Tolerance profile: Proportion of patients with no significant (grade ≥3 according to NCI CTCAE v4.03) toxicities responsible for irradiation breaks

SECONDARY OUTCOMES:
Quality of life measured by the EORTC QLQ-C30 (version 3.0) | From treatment start to 5 years after the end of radiotherapy
The acute and late toxicities assessed according to NCI CTCAE v4.03 | From treatment start to 5 years after the end of radiotherapy
The 6- and 12-month locoregional control rates defined by the proportion of patients with no local disease progression at 6 and 12 months after the end of radiotherapy | at 6 and 12 months after the end of radiotherapy
Duration of response defined by the time elapsed from first objective response to progression or death from any cause | From months 3 to progression
Quality of life measured by the additional colorectal module QLQ-CR 29 | From treatment start to 5 years after the end of radiotherapy
Quality of life measured by the Vaizey incontinence scale | From treatment start to 5 years after the end of radiotherapy
The acute and late toxicities assessed according the SOMA/LENT scale | From treatment start to 5 years after the end of radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Carmen FLORESCU, MD, Principal Investigator — Centre François Baclesse
Locations (8):
- France (8):
  - Institut de Cancérologie de l'Ouest - Centre Paul Papin, Angers
  - Centre François Baclesse, Caen
  - Centre Léon Berard, Lyon
  - Centre Antoine Lacassagne, Nice
  - Institut de cancérologie de l'Ouest, Saint-Herblain
  - Centre Paul Strauss, Strasbourg
  - IUCT-Oncopole, Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No